CLINICAL TRIAL: NCT01644682
Title: Replacement of Insecticides to Control Visceral Leishmaniasis
Brief Title: Replacement of Insecticides to Control Visceral Leishmaniasis (VL)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Rajendra Memorial Research Institute of Medical Sciences (Other); B.P. Koirala Institute of Health Sciences (Other); Directorate General of Health Services, GoB (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: PR-11045
Record Dates: First submitted 2012-07-17; First posted 2012-07-19 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2012-07

CONDITIONS: Cost-effective and Sustainable Vector Control Methods Will be Established to Reduce VL in India, Bangladesh and Nepal
Keywords: Visceral leishmaniasis; insecticide; wall lining; KO TAB123; Household; Kala-azar endemic area
MeSH Terms: conditions — Leishmaniasis, Visceral | interventions — Insecticides

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm-1 (Experimental): In each country, this arm constitute with 6 clusters where 2 from high, 2 from medium and 2 from low shadfly destiny. Each cluster has 50 households. It will receive IWFPL intervention.
  Interventions: Other: IWFPL
- Arm-2 (Experimental): In each country, this arm constitute with 6 clusters where 2 from high, 2 from medium and 2 from low shadfly destiny. Each cluster has 50 households. It will receive IDWL intervention.
  Interventions: Other: IDWL
- Arm-3 (Experimental): In each country, this arm constitute with 6 clusters where 2 from high, 2 from medium and 2 from low shadfly destiny. Each cluster has 50 households. It will receive ITN intervention.
  Interventions: Other: ITN
- Control (No Intervention): In each country, this arm constitute with 6 clusters where 2 from high, 2 from medium and 2 from low shadfly destiny. Each cluster has 50 households. It will not receive any intervention, Control group

INTERVENTIONS:
Other: IWFPL — Indoor house walls and floors will be plastered with lime (a traditional method known in the study areas) including treatment of outdoor breeding places with lime and bleaching powder to inhibit sandfly breeding
  Other Names: Insecticide
  Arms: Arm-1
Other: IDWL — Install durable wall lining containing deltamethrin to kill immature stage and as well as adult sand flies
  Other Names: Insecticide
  Arms: Arm-2
Other: ITN — Impregnation of existing bed-nets available in the community with slow release insecticide, deltamethrin
  Other Names: Insecticide
  Arms: Arm-3

SUMMARY:
Visceral leishmaniasis (VL) is a public health problem in Bangladesh, India and Nepal. To control the disease in these three countries a National kala-azar elimination program is ongoing. One of the major pillars of the elimination program is VL vector control. Currently there is a no public VL vector control program in Bangladesh. In India the program is depending on Indoor Residual Spraying with insecticides. IRS with DDT and in Nepal on Alpha-cypermethrin. The sand fly, vector of VL is already resistant to DDT and hurdles related with IRS i.e. funds, logistics and human resources make IRS unsustainable VL vector control method in Nepal. Thus alternative to IRS for VL vector control is highly desirable for the success of national kala-azar elimination program in these three countries.

Through current research activities we will compare the effectiveness of three effective VL vector control methods. They are 1) Plastering of household walls with lime (a traditional method known in the study areas),treatment of possible sand-fly breeding places with lime and bleaching powder; 2) Installing durable wall lining containing deltamethrin in the main living room(s) of households; 3) Impregnation of existing bed-nets with slow release insecticide tablet containing deltamethrin.

The study finding will be important for the national elimination program of the three countries through discovering the most effective VL vector control method.

DETAILED DESCRIPTION:
Visceral leishamniasis (VL; known as kala-azar in the Indian Sub-continent) is a deadly parasitic disease if left untreated. The disease is reported from 109 districts (Bangladesh-45, India-52 and Nepal-12). VL elimination programme was launched in 2005 between the three countries with the set target to reduce the cases one in 10,000 populations. Toward this set target, vector control will play a significant role. Based on the experiences in the past during malaria eradication period Indoor residual spraying (IRS) with insecticides is taken as the main pillar of VL vector control. Operation like IRS is expensive, labour-intensive, require sustainable infrastructures, supplies of insecticide, spraying equipment, trained personnel and funding over a long-term of period. These doubts about the sustainability of IRS in poor resource settings like Bangladesh. Thus alternative of IRS other vector control tool is highly desired. Current research activities will explore for the alternatives of IRS (here defined as "insecticide"). The proposed three different types of alternative of IRS are: 1) Plastering of household walls with lime (a traditional method known in the study areas), treatment of possible sand-fly breeding places with lime and bleaching powder; 2) Installing durable wall lining containing deltamethrin in the main living room(s) of households; 3) Impregnation of existing bed-nets with slow release insecticide tablet containing deltamethrin.

The study will include three different types of intervention arm and one control arm; Arm: 1) Indoor house walls and floors will be plastered with lime (a traditional method known in the study areas) including treatment of outdoor breeding places with lime and bleaching powder to inhibit sand fly breeding. Arm: 2) Installing of durable wall lining containing deltamethrin to kill immature stage of sand flies. Arm: 3) Impregnation of existing bed-nets with slow release insecticide, deltamethrin and 4) Control group, no intervention. VL endemic areas with 1200 households will be selected and identified 24 clusters based on geographic characteristics. Minimum distance between each cluster will be about 50 meters. Each cluster will have 50 households (HHs) where the different interventions will be applied. Five HHs will be selected randomly from each cluster to measure the intervention effect on sandfly density on 2 consecutive nights using CDC light traps at 4, 12, 24 and 52 weeks after intervention. Baseline sand fly densities will be measured at 2 weeks before introducing the intervention. Based on base line sandfly data the clusters will be ranked as high, moderate and low and from them equal number of clusters will be assigned for each intervention arm as well as control arm. Control HHs will receive commercial insecticide treated bed-nets after the study is over. This study will be a multi-centre cluster randomized trial with three vector control methods and will be carried out in ICDDR,B, Bangladesh, RMRI, India and in BPKIHS, Dahran, Nepal simultaneously during a 12 months period. A total of 3600 households in the three countries (Bangladesh-1200, India-1200 and Nepal-1200 HHs) will be included in the study.

The cost of interventions will be assessed applying a combination of bottom-up and top-down costing approach from the provider's perspective only. Costs attributable to effectiveness of the interventions (i.e. reduction of sandfly density by intervention) will be calculated separately for comparison among three types of intervention. Firstly; all inputs to be mobilized for implementing each of the intervention will be identified, quantified and valued in local currency separately. Based on the relationship of the inputs to outputs, costs will be broadly classified into fixed cost and variable cost. Standard procedure will be followed for annualization of capital costs using replacement cost, useful lifetime, discounting rate and corresponding annualization factor taken from the standard table.

Shadow pricing will be considered for inputs to be donated for the study purpose by partner agencies. Allocation factors (e.g. % time spent by staff, % used etc) will be applied to apportion joint costs. Summing-up the fixed and variable costs over all total cost of each intervention will be calculated separately. Average or unit cost will be calculated dividing total cost of each intervention by the corresponding number of households that received the intervention. Finally relationship between cost and effectiveness of corresponding intervention(s) will be represented by cost and effectiveness ratio for comparison.

ELIGIBILITY:
Inclusion Criteria:

* Household head who agree to participate in the study

Exclusion Criteria:

* Household head who does not agree to participate in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3600 (Actual)
Dates: Start 2012-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Measurement of efficacy of interventions | 12 months
  Efficacy will be measured by the reduction of sand-fly density by intervention compared to control measured by sand-fly density at 4 weeks, 12 weeks, 24 weeks and 12 months after intervention; percentage mortality of sand-fly assessed by WHO Cone Bioassay test on wall and impregnated net compared to control at 4 weeks, 12 weeks, 24 weeks and 12 months after intervention.

SECONDARY OUTCOMES:
Estimation of intervention costs and its acceptability | 12 months
  Fixed costs (equipment/accessories, apportioned staff salary, non-recurrent training, social mobilization etc.) and variable costs (lime, bleaching powder, K0 tab 123, wall lining, labor charge, transportation, travel cost etc.) data will be collected through projects financial database, household level inventory that received intervention(s), key informant interview with field supervisors/technicians, and record review. Relationship between cost and effectiveness of corresponding intervention(s) will be represented by cost and effectiveness ratio for comparison.
  Acceptability survey will be carried out through structure questionnaire in all the experimental arms. The survey will be conducted at 6 weeks after intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Godagari, Rajshahi, Bangladesh